CLINICAL TRIAL: NCT06674876
Title: WINGS Project: Wellness Interventions for Nurses' Post Traumatic Growth and Self Care : A Pilot Randomized Controlled Trial Study
Brief Title: Wellness Intervention for Nurses Post Traumatic Growth and Selfcare
Acronym: WINGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: University of East London (Other); Kennesaw State University (Other)
Responsible Party: Principal Investigator, Nasreen Lalani, PhD, MSN, RN, Assistant Professor, Purdue University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-1156
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Trauma, Psychological; Moral Injury; Compassion Fatigue
Keywords: resilience; trauma; nurses; palliative care; subjective wellbeing; post traumatic growth; self reflexivity; existential wellbeing; blog writing
MeSH Terms: conditions — Psychological Trauma; Stress Disorders, Post-Traumatic; Compassion Fatigue; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Palliative care nurses who participated in Presurvey were then divided under one control and two intervention groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): This group only filled pre and post surveys at baseline, 4 and 6 weeks
- IG 1-Blog writing (Other): This group were asked to write 2blogs a week for four weeks based on SOPHIE framework
  Interventions: Behavioral: Blog writing
- IG2-Blog writing and workshop (Other): This group was asked to write 2bolgs a week for four weeks and then attend a 4hour wellness workshop
  Interventions: Behavioral: Blog writing

INTERVENTIONS:
Behavioral: Blog writing — Participants were asked to write 2blogs online for four weeks and attend a 4hours wellness workshop
  Other Names: wellness workshop
  Arms: IG 1-Blog writing; IG2-Blog writing and workshop

SUMMARY:
Nurses working in home and hospice care settings find their roles emotionally challenging and are at high risk for trauma, strain and fatigue. Such sufferings were high among nurses during the Covid-19 pandemic. Our study tested the effectiveness of a self-reflexive wellness intervention to promote resilience, posttraumatic growth and subjective wellbeing among nurses. Participants were divided in three different groups. One group did not intervention whereas the other two were assigned writing 2 blogs each week and attending a wellness workshop. Findings showed that writing weekly blogs helped nurses to be self reflexive about their feelings, generated self-awareness and improved their wellbeing.

DETAILED DESCRIPTION:
Recent pandemic crisis has further exposed nurses to added vulnerabilities, trauma, and sufferings including increased burnouts, suicide rates, psychological and existential crisis. Nurses working in nursing homes, long term care and hospice settings require increased support to embrace reappraise their trauma and suffering in order to gain personal strength and growth. Our study aimed to examine the effectiveness of 'SOPHIE' (Self-exploration through Ontological, Phenomenological, and Humanistic, Ideological, and Existential expressions) as a self-reflective wellness intervention to promote resilience, posttraumatic growth, and subjective wellbeing among nurses working in the palliative care settings.

The specific aims of the study included: 1) To determine the extent of self-perceived trauma, resilience, and subjective wellbeing among nurses working in palliative care settings (i.e., nursing homes, hospice, and long-term care facilities) 2) To identify associated factors contributing to trauma, resilience, and subjective wellbeing of nurses. 3) To evaluate the effectiveness of a self-reflective wellness intervention tool in promoting fostering resilience, posttraumatic growth, and subjective wellbeing of nurses. The study was guided by NPT (Nurse Psychological Trauma) and SOHIE framework. Using a quasi-experimental Pre and Posttest design, we enrolled 160 participants in the study. Participants in the intervention group were asked to write 2 blogs every week online using Qualtrics and attend a 4 hour wellness workshop. Pre- and post-intervention surveys were sent online at the baseline, four weeks, and six weeks following intervention.

Pre and post-test surveys were analyzed using the SPSS, a quantitative statistical tool and included self-reported outcomes measures of post traumatic growth, resilience and subjective wellbeing between the control and intervention groups at baseline, 4 weeks and 6 weeks of the study. Demographic data was also analyzed. The participant characteristics include participant's age, gender, level of education, position, training. whereas research outcome variables include post traumatic growth, resilience, and subjective wellbeing. Inferential statistics was used to test the hypothesis under the study. Statistical significance kept at p<0.05 (two-sided) level. Content analysis was done for the descriptive data in the survey including blogs and feedback regarding the intervention. Weekly blogs received were analyzed using thematic analysis approach.

Findings showed significant differences in subjective wellbeing of nurses post intervention. Nearly all participants found blog writing as a supportive and therapeutic intervention that helped them to reflect on their experiences of anxiety, trauma and distress.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are actively practicing as registered nurses in palliative care settings (i.e., nursing homes, hospices, and long-term care settings); 2) individuals who can read and speak English, and 3) individuals who are age 18 years or above.

Exclusion Criteria:

* Those who are not registered nurses and are not working in palliative care setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Resilience | at baseline, 4 and 6 weeks
  Resilience is defined as ability to adapt. it was measured using Brief resilience scale
Subjective wellbeing | at baseline, 4 and 6 weeks
  Measured using Subjective Wellbeing Inventory (SUBI) scale
Post traumatic growth | at baseline, 4 and 6 weeks
  measured using Posttraumatic Growth Inventory (PTGI) Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nasreen Lalani, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No